CLINICAL TRIAL: NCT05033925
Title: Safety and Clinical Efficacy Evaluation of Awar-awar Leaves (Ficus Septica Burm. F.) Active Fraction Capsule as Chemotherapy Complement in Stage IV Breast Cancer Patients
Brief Title: Ficus Septica Leaves Fraction as a Complementary Therapy for Stadium IV Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Ahmad Dahlan University (Unknown); Dr. Kariadi General Hospital (Unknown); PT Konimex (Unknown); LPDP, Kementerian Keuangan, Indonesia (Unknown)
Responsible Party: Principal Investigator, Nanang Fakhrudin, Head of Department of Pharmaceutical Biology, Faculty of Pharmacy, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UKFC-PU-2019-01-08; PRJ-82/LPDP/2019 (Other Grant/Funding Number: Lembaga Pengelola Dana Pendidikan, Kemenkeu, Indonesia)
Record Dates: First submitted 2021-08-05; First posted 2021-09-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Stage IV
Keywords: ficus septica; cancer; doxorubicin; adjuvant
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind; Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): receive a plasebo capsule 2 doses per day
  Interventions: Other: Placebo capsule
- FADA 800 mg/day (Experimental): receive FADA capsules twice a day (each 400 mg)
  Interventions: Dietary Supplement: FADA (active fraction of Ficus septica leaf) 800 mg/day
- FADA 2000 mg/day (Experimental): receive FADA capsules twice a day (each 1000 mg)
  Interventions: Dietary Supplement: FADA (active fraction of Ficus septica leaf) 2000 mg/day

INTERVENTIONS:
Dietary Supplement: FADA (active fraction of Ficus septica leaf) 800 mg/day — FADA is given twice a day (total dose of 800 per day per patient)
  Arms: FADA 800 mg/day
Dietary Supplement: FADA (active fraction of Ficus septica leaf) 2000 mg/day — FADA is given twice a day (total dose of 2000 per day per patient)
  Arms: FADA 2000 mg/day
Other: Placebo capsule — Placebo capsule is given twice a day
  Arms: Placebo

SUMMARY:
The purpose of this research is to assess the safety profile and clinical benefit of Awar-Awar leaf active fraction as a complementary therapy in chemotherapy of stage IV breast cancer

DETAILED DESCRIPTION:
The study uses a double blind design and randomized controlled trial that compares the safety and clinical efficacy profiles of 3 treatment groups (each consists of 97 subjects who received chemotherapy for 6 cycles). The treatment group was given FADA at a dose of 800 mg/day and 2000 mg/day compared to the placebo group. Interim analysis is carried out after 25% of the subjects completed 3 cycles of chemotherapy; whereas interim analysis II is carried out after 50% of the subjects completed 3 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female, at least 18 years old
* Welfare scale 0, 1, and 2 (ECOG - WHO)
* Patients with stage IV breast cancer who have histopathological data according to the TNM Classification of Malignant Tumors (TNM) from American Joint Committee on Cancer (AJCC) 8th edition 2017
* Patients who are willing to participate in the test and sign an informed consent
* Patients who undergo breast cancer chemotherapy with luminal B sub-type or triple negative with anthracycline base
* Patients who are willing and able to fill out a questionnaire
* The patients who are willing and able to comply with the test protocols during the test

Exclusion Criteria:

* Unable to meet the test protocol
* Patients with liver and kidney disorders
* Patients with other diseases/disorders that are meaningful according to the investigators will be excluded from the test
* Patients with cancer that has metastasized to the brain
* Pregnant women and breastfeeding mothers
* Patients with the ejection fraction smaller-than or equal to 55%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment | The measurement is at 3-7 days before the 4th cycle of chemotherapy (each cycle is 21 days), and 14-21 days after the 6th cycle (each cycle is 21 days)
  The change of quality of life index during 6 cycles of chemotherapy (each cycle is 21 days). The score ranges from 0 (best) to 100 (worst).

SECONDARY OUTCOMES:
Adverse events (AEs) and Serious Adverse Events (SAEs). | throughout the duration of the trial (126 days) or 6 cycles of chemotherapy (each cycle is 21 days)
  Safety data will be collected by monitoring and recording all adverse events (AEs) and Serious Adverse Events(SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: dr. Santosa, Ph.D, Principal Investigator — Dr. Kariadi General Hospital
Locations (1):
- Dr. Kariadi General Hospital, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No